CLINICAL TRIAL: NCT01524601
Title: The RITA-study -- An Open Study to Evaluate the Blood Lipid Lowering Effect of Rosuvastatin Versus Fluvastatin and the Bilateral Interaction Between Everolimus and Rosuvastatin in Renal Transplant Recipients
Brief Title: The Rosuvastatin In TrAnsplant Recipients Study
Acronym: RITA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo School of Pharmacy (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RITA-11
Record Dates: First submitted 2012-01-24; First posted 2012-02-02 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Disorder Related to Renal Transplantation; Hypercholesterolemia
Keywords: Immunosuppression; Everolimus; rosuvastatin; fluvastatin; Lipid lowering
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rosuvastatin (Experimental): Rosuvastatin treatment for 4 weeks
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — 20 mg rosuvastatin for 4 weeks
  Other Names: Crestor

SUMMARY:
Renal transplant recipients need life long immunosuppression and one of the new drugs is everolimus. Everolimus is a potent immunosuppressive drug and one of the main side-effects are increased blood cholesterol levels. Many renal transplant recipients are treated with a cholesterol lowering agent, mainly fluvastatin. Rosuvastatin is a new cholesterol lowering drug on the market with a potential higher cholesterol lowering potency. In the present study the investigators will examine the hypothesis that rosuvastatin reduce cholesterol levels more than fluvastatin in renal transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients with stable renal function (plasma creatinine < 200 µmol/L)
* Renal transplant recipients on an everolimus and fluvastatin based therapy for minimum 3 months prior to inclusion
* > 18 years of age
* Male patient or female patient without childbearing potential (surgically sterilized or postmenopausal) or if female of childbearing potential; is not lactating, has a negative pregnancy test at screening and is willing to utilize an effective method of contraception throughout the study period and for 90 days following discontinuation of the study drugs
* Signed informed consent

Exclusion Criteria:

* Patients experiencing an acute rejection episode within 2 weeks before or after inclusion, whether proven by biopsy or not
* Patients with a known hypersensitivity to rosuvastatin
* Change in enzyme inducing or inhibiting drugs within the last 2 weeks prior to and throughout the study [e.g. barbiturates, rifampicin, ketoconazole, erythromycin, cimetidine and similar drugs]
* Pregnant or nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
compare the treatment efficacy (blood lipid lowering effect) of rosuvastatin versus fluvastatin | 4 weeks
  Compare the blood lipid levels before and after switch from fluvastatin to rosuvastatin
Area Under Curve (AUC) of rosuvastatin in renal transplant recipients treated with everolimus. Time frame: predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post dose. | 4 weeks
  Compare 24-h pharmacokinetics of renal transplant recipients with historic controls

SECONDARY OUTCOMES:
1. Area Under Curve (AUC) of everolimus during rosuvastatin versus fluvastatin therapy, including intracellular everolimus concentrations within T-lymphocytes. Time frame: predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours post-dose. | 4 weeks
2. Investigate P-gp activity in whole blood in everolimus treated patients | 4 weeks
3. Study inter individual variation in rosuvastatin and everolimus pharmacokinetics in renal transplant recipients due to polymorphism in the genes encoding P-gp, OATP1B1 and CYP3A5 | 4 weeks
4. Compare effect of rosuvastatin versus fluvastatin therapy on the renal function (eGFR) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anders Åsberg, PhD, Study Director — University of Oslo
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Norway

REFERENCES:
- [Derived] Robertsen I, Asberg A, Granseth T, Vethe NT, Akhlaghi F, Ghareeb M, Molden E, Reier-Nilsen M, Holdaas H, Midtvedt K. More potent lipid-lowering effect by rosuvastatin compared with fluvastatin in everolimus-treated renal transplant recipients. Transplantation. 2014 Jun 27;97(12):1266-71. doi: 10.1097/01.TP.0000443225.66960.7e. PMID 24521776